CLINICAL TRIAL: NCT01001663
Title: Comparison of the FemoSeal® Arterial Closure Device to Manual Compression After Coronary Angiography: the CLOSE-UP I Randomized Trial
Brief Title: Comparison of the FemoSeal® Arterial Closure Device to Manual Compression After Coronary Angiography
Acronym: CLOSE-UP I
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Vingmed Danmark A/S (Individual)
Responsible Party: Principal Investigator, Evald Hoej Christiansen, MD, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-20090101
Record Dates: First submitted 2009-10-16; First posted 2009-10-26 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Coronary Angiography Via Femoral Artery Access
Keywords: CAG

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FemoSeal® (Experimental): Closure device for femoral artery access closure
  Interventions: Device: FemoSeal®
- Manual compression (Active Comparator): Conventional manual compression
  Interventions: Other: Manual compression

INTERVENTIONS:
Device: FemoSeal® — Closure device for femoral artery access closure
  Arms: FemoSeal®
Other: Manual compression — Conventional manual compression
  Arms: Manual compression

SUMMARY:
Is the FemoSeal® closure device safer and more comfortable than manual compression for femoral artery access closure after coronary angiography?

DETAILED DESCRIPTION:
Access site complication after coronary angiography is still a challenge in everyday practice. The FemoSeal® closure device has proven very safe as shown in the swedish SCAAR registry. This study is aimed to investigate, in a randomized design, if the FemoSeal® has an advantage in safety and efficacy over manual compression.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be at least 18 years old
* Patients undergoing femoral access coronary angiography
* Patient must be competent for providing informed, written consent
* Only 6F sheath

Exclusion Criteria:

* Percutaneous coronary intervention
* Intra coronary measurements (FFR, IVUS, OCT, NIR)
* Groin hematoma before closure
* Pseudoaneurysm or AV fistula
* Significant stenosis of ilial or femoral artery
* Prior peripheral artery surgery
* INR > 3,0
* Platelet count < 120 million per millilitre blood
* Coagulopathy (bleeding disorder)
* Thrombolysis in the last 24h
* Planned heparin infusion after the procedure
* Pregnancy
* Uncontrolled hypertension > 200 mmHg / 110 mmHg
* Femoral access device closure in the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1005 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Rate of ipsilateral palpable groin hematomas with largest diameter exceeding 5 cm. | 20 minutes, 1 hour and at discharge, pooled

SECONDARY OUTCOMES:
Rate of ipsilateral palpable groin hematomas with largest diameter exceeding 5 cm. Patient self-measurements. | 14 days
Composite of: major vascular complications necessitating surgical repair, A-V fistulation, pseudoaneurysm needing treatment, major bleeding needing transfusion and infection needing antibiotics . | 14 days
Time to hemostasis, from sheath removal to hemostasis is achieved | 14 days
Time from end of closure procedure to ambulation. 1h bedrest recommended. | 14 days
Device deployment failure | 20 minutes
Time to cessation of continuous minor oozing measured from the end of the closure procedure | 14 days
Need for repeated manual compression after end of the closure procedure | 14 days
Pain and discomfort measured on a numerical pain rating scale (0-10) | 20 min
Vasovagal reaction (clinical signs AND Systolic BP drop of more than 30 mmHg AND/OR pulse drop more than 30 b/min. AND reversible immediately after treatment by atropin, fluids) | 20 minutes
The patient seeking medical assistance for all-cause closure site related symptoms after discharge. | 14 days
Pain and discomfort measured on a numerical pain rating scale (0-10) | 1 hour
Pain and discomfort measured on a numerical pain rating scale (0-10) | Discharge
Pain and discomfort measured on a numerical pain rating scale (0-10) | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Niels R. Holm, MD, Principal Investigator — Aarhus University Hospital Skejby
Locations (1):
- Aarhus University Hospital Skejby, Aarhus N, Denmark

REFERENCES:
- [Derived] Holm NR, Sindberg B, Schou M, Maeng M, Kaltoft A, Bottcher M, Krusell LR, Hjort J, Thuesen L, Terkelsen CJ, Christiansen EH, Botker HE, Kristensen SD, Lassen JF; CLOSE-UP study group. Randomised comparison of manual compression and FemoSeal vascular closure device for closure after femoral artery access coronary angiography: the CLOSure dEvices Used in everyday Practice (CLOSE-UP) study. EuroIntervention. 2014 Jun;10(2):183-90. doi: 10.4244/EIJV10I2A31. PMID 24603054
- [Derived] Sindberg B, Schou M, Hansen L, Christiansen KJ, Jorgensen KS, Soltoft M, Holm NR, Maeng M, Kristensen SD, Lassen JF. Pain and discomfort in closure of femoral access coronary angiography. The CLOSuredEvices Used in everyday Practice (CLOSE-UP) pain sub study. Eur J Cardiovasc Nurs. 2014 Jun;13(3):221-6. doi: 10.1177/1474515113482809. Epub 2013 Mar 25. PMID 23532433